CLINICAL TRIAL: NCT04341948
Title: Treatment of Post-Operative Pain Following Orthopedic Surgery With SPRINT® Peripheral Nerve Stimulation (PNS) System in a Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Treatment of Post-Operative Pain Following Orthopedic Surgery With SPRINT® Peripheral Nerve Stimulation (PNS) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPR Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0150-CSP-000; CDMRP-OR170165 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain; Total Knee Replacement; Total Knee Arthroplasty; Partial Knee Replacement
Keywords: Pain, Postoperative; Musculoskeletal Diseases; Postoperative Complications; Nervous System Diseases; Pain; Neurologic Manifestations; Signs and Symptoms
MeSH Terms: conditions — Pain, Postoperative; Musculoskeletal Diseases; Postoperative Complications; Nervous System Diseases; Pain; Neurologic Manifestations; Signs and Symptoms | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Treatment) (Active Comparator): Participants in Group 1 will have Leads placed by the nerves of the mid to upper thigh. These participants will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and will receive electrical stimulation for 8 weeks.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System
- Group 2 (Control) (Sham Comparator): Participants in Group 2 will have Leads placed by the nerves of the mid to upper thigh. These participants will then use the SPRINT Peripheral Nerve Stimulation (PNS) System and receive 8 weeks of sham stimulation. Participants will then have the option to crossover and receive stimulation therapy.
  Interventions: Device: SPRINT Peripheral Nerve Stimulation (PNS) System

INTERVENTIONS:
Device: SPRINT Peripheral Nerve Stimulation (PNS) System — The SPRINT System delivers mild electrical stimulation to nerves in the affected limb. The SPRINT System includes two small wires (called "Leads") that are placed through the skin in the upper leg. It also includes a device worn on the body that delivers stimulation (called the SPRINT Stimulator).
  Other Names: SPRINT; SPRINT System

SUMMARY:
The purpose of this study is to gather information about how knee pain changes when small amounts of electricity are delivered to the nerves in the leg. This study will involve the use of a Peripheral Nerve Stimulation (PNS) System that is made by SPR Therapeutics (the sponsor of the study). The SPRINT PNS System was cleared by the FDA for up to 60 days of use in the back and/or extremities for the management of acute and chronic pain.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 21 years old
* Underwent a 1. primary total knee replacement (TKR), 2. secondary/revision TKR or 3. Partial/unicompartmental knee replacement (PKR)
* Knee pain directly resulting from Knee Replacement surgery in affected knee

Key Exclusion Criteria:

* Current high opioid use
* Body Mass Index (BMI) > 40 kg/m2
* Conditions with increased risk of infection
* Implanted electronic device
* History of bleeding or clotting disorder.
* Uncontrolled Diabetes Mellitus Types I or II
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, San Diego, California
  - The Orthopaedic Institute, Gainesville, Florida
  - Better Health Clinical Research, Inc, Newnan, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Ali K. Valimahomed MD PLLC, Holmdel, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining informed consent, participants were evaluated for eligibility.
Groups:
- Group 1 (Treatment): Participants in Group 1 were consented and met all eligibility criteria prior to randomization. These participants had leads placed in their mid to upper thigh and received electrical stimulation for up to 8 weeks with the SPRINT Peripheral Nerve Stimulation (PNS) System.
- Group 2 (Control): Participants in Group 2 were consented and met all eligibility criteria prior to randomization. These participants had leads placed in their mid to upper thigh and received up to 8 weeks of sham stimulation. Three months after start of sham treatment, participants were given the option to crossover and receive electrical stimulation treatment with the SPRINT Peripheral Nerve Stimulation (PNS) System.
Period: Overall Study
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Started | 29 | 27
Randomized (All participants who were consented, met eligibility criteria, and were randomized.) | 29 | 27
Safety Analysis Set (All participants who were consented, randomized, and lead placement procedures attempted.) | 28 | 27
Full Analysis Set (Includes participants who were consented, randomized, continued to meet eligibility criteria prior to undergoing lead placement, and have data available for at least 1 lead during weeks 5-8 post-start of treatment (SOT). Participants who had a partial knee replacement or a revision knee replacement (enrolled only for exploratory analysis) are excluded.) | 20 | 21
Per Protocol Set (Includes participants who were consented, randomized, continued to meet eligibility criteria prior to lead placement, have data for at least 1 lead during weeks 5-8 post-start of treatment (SOT), reported coverage of sensations in the target areas during weeks 5-8 post-SOT (Group 1 only), have adequate diary completion, and continued study eligibility through the treatment period. Participants with partial or revision knee replacement (enrolled only for exploratory analysis) are excluded.) | 16 | 19
Group 2 Crossover Safety Set (Participants who were consented, randomized to Group 2 (Control), received sham stimulation treatment, and crossed over to receive electrical stimulation via the SPRINT Peripheral Nerve Stimulation (PNS) System.) | 0 | 11
Completed | 15 | 20
Not Completed | 14 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Participant | 6 | 3
Not completed — Lack of compliance by Participant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Treatment) | Group 2 (Control) | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.5) | 62.2 (7.6) | 63.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 27 | 27 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 17 | 22 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 27 | 56
Employment Status [Count of Participants; unit: Participants]
  Currently Working | 6 | 11 | 17
  Retired (not due to health) | 13 | 8 | 21
  Unemployed | 3 | 2 | 5
  Disabled / Retired (due to health) | 7 | 5 | 12
  Other (Retired (not due to health) and employed part-time) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Average Pain Intensity: Number of Participants With ≥ 50% Reduction in Average Pain Intensity
Description: All participants were asked to complete daily diaries to record their average knee pain during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain scores were calculated across the 7-day diary(s) at baseline and across weeks 5 to 8 post-start of treatment. Percent reduction was then calculated for each participant. To be considered a success, participants must have experienced ≥ 50% reduction in average knee pain. The number of successes is presented.
Time Frame: Baseline and 5 to 8 weeks post-Start of Treatment (SOT)
Population: Full Analysis Set presented. To account for missing data due to missed visits and early terminations, data were also imputed using a mixed-effects model.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
Participants | 12 | 5

2. Primary Outcome: Study-Related Adverse Device Effects
Description: At each study visit following the baseline assessment at Visit 1, participants were questioned if any changes in their medical status or condition have occurred since their previous visit. If the participant experienced a change that was a study-related adverse event, an Adverse Event Form was completed by the site. The number of participants that experienced at least one study-related adverse event is reported here. Adverse Events are reported by the trial phase in which they occurred: Group 1 Treatment (active stimulation), Group 2 Control (sham stimulation), and Group 2 Crossover Safety Set (active stimulation).
Time Frame: Up to 13 months for each Group 1 participant and up to 16 months for Group 2 participants that opted to cross over (time from baseline to last study visit)
Population: Safety Analysis Set presented.
Measure: Count of Participants; unit: Participants
Groups:
- Group 2 Crossover Safety Set: Participants who were consented, randomized to Group 2 (Control), received sham stimulation treatment, and crossed over to receive electrical stimulation via the SPRINT Peripheral Nerve Stimulation (PNS) System.
Arm/Group | Group 1 (Treatment) | Group 2 (Control) | Group 2 Crossover Safety Set
Number analyzed (Participants) | 28 | 27 | 11
Participants | 9 | 14 | 5

3. Secondary Outcome: Reduction in Average Pain Intensity: Number of Participants With ≥ 50% Reduction in Average Pain Intensity
Description: All participants were asked to complete daily diaries to record their average knee pain intensity during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain score was calculated across the 7-day diary(s) at baseline and across weeks 1 to 4 post-start of treatment. Percent reduction was then calculated for each participant. To be considered a success, participants must have experienced ≥ 50% reduction in average knee pain. The number of successes is presented.
Time Frame: Baseline and 1 to 4-weeks post-start of treatment (SOT)
Population: Full Analysis Set presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
Participants | 7 | 3

4. Secondary Outcome: Long-term Durability of Average Pain Relief: Number of Participants With ≥ 50% Reduction in Average Pain Intensity
Description: All participants were asked to complete daily diaries to record their average knee pain intensity during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The average pain score was calculated across the 7-day diary for each participant at baseline and at 3-, 6-, 9-, and 12-months post-start of treatment. Percent reduction was then calculated for each participant. To be considered a success, participants must have experienced ≥ 50% reduction in average knee pain. The number of successes is presented.
Time Frame: Baseline, 3-months post-start of treatment (SOT), 6-months post-SOT, 9-months post-SOT, 12-months post-SOT
Population: Full Analysis Set presented. According to the planned study protocol, Group 2 was not assessed for this outcome at 6, 9, and 12-months due to crossover to receive active stimulation. To account for missing data due to missed visits and early terminations, data were also imputed using a mixed-effects model for Group 2 at 3-months post-SOT and for Group 1 at 6, 9, and 12-months post-SOT.
Measure: Number; unit: participants (with imputed values)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
participants (with imputed values)
  3-months Post-SOT | 10.00 | 5.00
  6-months Post-SOT: number analyzed (Participants) | 20 | 0
  6-months Post-SOT | 9.96 |
  9-months Post-SOT: number analyzed (Participants) | 20 | 0
  9-months Post-SOT | 9.02 |
  12-months Post-SOT: number analyzed (Participants) | 20 | 0
  12-months Post-SOT | 10.36 |

5. Secondary Outcome: Mean Pain Relief
Description: All participants were asked to complete daily diaries to record their average knee pain intensity during the past 24 hours on each day of a 7-day period using an 11-point numerical rating scale where 0 represents "No Pain" and 10 represents "Pain as bad as you can imagine." The mean pain score was calculated across the 7-day diary(s) for each participant at baseline, 1-4 weeks post-start of treatment (SOT), 5-8 weeks post-SOT, and at 3-, 6-, 9-, and 12-months post-SOT. The mean pain score is presented.
Time Frame: Baseline, 1 to 4-weeks post-start of treatment (SOT), 5 to 8-weeks post-SOT, 3-months post-SOT, 6-months post-SOT, 9-months post-SOT, and 12-months post-SOT
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale (with imputed values)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
score on a scale (with imputed values)
  Baseline | 7.26 (1.24) | 7.21 (1.44)
  1 to 4 weeks Post-SOT | 4.37 (2.02) | 5.65 (2.16)
  5 to 8 weeks Post-SOT | 3.32 (2.18) | 5.34 (2.56)
  3-months Post-SOT | 3.69 (2.67) | 5.37 (2.76)
  6-months Post-SOT: number analyzed (Participants) | 20 | 0
  6-months Post-SOT | 4.04 (2.78) |
  9-months Post-SOT: number analyzed (Participants) | 20 | 0
  9-months Post-SOT | 4.00 (2.71) |
  12-months Post-SOT: number analyzed (Participants) | 20 | 0
  12-months Post-SOT | 4.15 (2.75) |

6. Secondary Outcome: Pain Medication Usage
Description: Participants recorded the amount/type of analgesics used in daily diaries. A blinded, third-party medication committee reviewed participants' diary medications for each time period to determine if each participant's analgesic usage changed. The committee determined whether there was No change (no change in dosage or change is not clinically meaningful to impact pain outcomes), an Increase (clinically meaningful increase in medication that would impact pain outcomes), or a Decrease (clinically meaningful decrease in medication that would impact pain outcomes) for each time period compared to baseline. The number of participants with a Decrease in analgesic medication usage for pain are reported. Participants that did not report any pain medications during the study were excluded from the analysis.
Time Frame: Baseline, 1 to 4 weeks post-start of treatment (SOT), and 5 to 8 weeks post-SOT, 3-months post-SOT, 6-months post-SOT, 9-months post-SOT, and 12-months post-SOT
Population: Full Analysis Set presented. According to the planned study protocol, Group 2 was not assessed for this outcome at 6, 9, and 12-months due to crossover to receive active stimulation. Participants that did not report any pain medications during the study were excluded. Data were not available for one Group 2 participant at 3-months post-SOT, five Group 1 participants at 6-months post-SOT, three Group 1 participants at 9-months post-SOT, and six Group 1 participants at 12-months post-SOT.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 17 | 20
Participants
  1 to 4 weeks post-SOT | 8 | 9
  5 to 8 weeks post-SOT | 11 | 10
  3-months post-SOT: number analyzed (Participants) | 17 | 19
  3-months post-SOT | 8 | 8
  6-months post-SOT: number analyzed (Participants) | 12 | 0
  6-months post-SOT | 5 |
  9-months post-SOT: number analyzed (Participants) | 14 | 0
  9-months post-SOT | 4 |
  12-months post-SOT: number analyzed (Participants) | 11 | 0
  12-months post-SOT | 4 |

7. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) questionnaire has 13 questions that assess rumination, magnification, and helplessness. Participants are asked to think back on painful experiences in the past and reflect on how often they had specific thoughts or feelings. Each of the 13 questions is scored on a 5-point scale where 0 represents "not at all," and 4 represents "all the time." The scores from each question were summed for each participant to provide a total PCS score, with a possible range from 0 to 52 with higher scores indicating a greater tendency to catastrophize pain (i.e. a higher score indicates a worse outcome). The mean score for each time point is presented.
Time Frame: Baseline (Visit 1), 4-weeks post-SOT (Visit 6), and 8-weeks post-SOT (Visit 10)
Population: Full Analysis Set presented. Data were not available for one Group 1 participant and two Group 2 participants at 4-weeks post-SOT and for one Group 2 participant at 8-weeks post-SOT.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
score on a scale
  Visit 1: Baseline | 24.30 (12.92) | 27.14 (16.81)
  Visit 6: 4-weeks Post-SOT: number analyzed (Participants) | 19 | 19
  Visit 6: 4-weeks Post-SOT | 12.53 (11.41) | 16.47 (14.63)
  Visit 10: 8-weeks Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 10: 8-weeks Post-SOT | 9.30 (8.29) | 14.75 (14.35)

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change (PGIC) Survey asks participants to rate their improvement with treatment on a 7-point scale ranging from -3 to 0 to +3, where -3 represents "very much worse," 0 is "no change," and +3 represents "very much improved" as compared to before stimulation treatment. The participants combine all the components of their experience into one overall score. The mean score of each group was calculated for each time frame.
Time Frame: 4-weeks post-start of treatment (SOT)(Visit 6), 8-weeks post-SOT (Visit 10), 3-months post-SOT (Visit 11), 6-months post-SOT (Visit 12), 9-months post-SOT (Visit 13), and 12-months post-SOT (Visit 14)
Population: Full Analysis Set presented. According to the planned study protocol, Group 2 was not assessed for this outcome at 6, 9, and 12-months due to crossover to receive active stimulation. Missing data due to missed visits and early terminations were also imputed using a mixed-effects model for outcomes at 6, 9, and 12-months post-SOT. Data were not available for one Group 1 and two Group 2 participants at 4-weeks, one Group 2 participant at 8-weeks, and one Group 2 participant at 3-months post-SOT.
Measure: Mean (Standard Deviation); unit: score on a scale (with imputed values)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
score on a scale (with imputed values)
  Visit 6: 4-weeks Post-SOT: number analyzed (Participants) | 19 | 19
  Visit 6: 4-weeks Post-SOT | 1.42 (1.22) | 1.05 (0.97)
  Visit 10: 8-weeks Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 10: 8-weeks Post-SOT | 1.80 (1.06) | 1.15 (1.18)
  Visit 11: 3-months Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 11: 3-months Post-SOT | 1.75 (1.16) | 0.75 (1.25)
  Visit 12: 6-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 12: 6-months Post-SOT | 1.32 (1.49) |
  Visit 13: 9-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 13: 9-months Post-SOT | 1.01 (1.58) |
  Visit 14: 12-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 14: 12-months Post-SOT | 1.11 (1.36) |

9. Secondary Outcome: Pain Interference: Number of Participants With ≥ 50% Reduction in Pain Interference
Description: Question 9 of the Brief Pain Inventory-Short Form (BPI-9) is a 7-part question that assesses the level of interference that participants experience in their daily lives due to pain. The 7 categories are general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Participants were asked to rate how much their post-surgical knee pain interferes with each aspect on an 11-point numerical scale where 0 represents "Does Not Interfere" and 10 represents "Completely Interferes." The average of these 7 scores was calculated for each participant at each time point. Percent reduction was then calculated for each participant. To be considered a success, participants must have experienced ≥ 50% reduction in pain interference. The number of successes is presented.
Time Frame: Baseline (Visit 1), 8-weeks post-start of treatment (SOT) (Visit 10), 3-months post-SOT (Visit 11), 6-months post-SOT (Visit 12), 9-months post-SOT (Visit 13), and 12-months post-SOT (Visit 14)
Population: Full Analysis Set presented. According to the planned study protocol, Group 2 was not assessed for this outcome at 6, 9, and 12-months due to crossover to receive active stimulation. For participants that completed treatment, missing data due to missed visits and early terminations were also imputed using a mixed-effects model at 6, 9, and 12-months post-SOT. Data were not available for one Group 2 participant at 8-weeks and 3-months post-SOT.
Measure: Number; unit: participants (with imputed values)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
participants (with imputed values)
  Visit 10: 8-weeks Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 10: 8-weeks Post-SOT | 13.00 | 11.00
  Visit 11: 3-months Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 11: 3-months Post-SOT | 11.00 | 6.00
  Visit 12: 6-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 12: 6-months Post-SOT | 11.20 |
  Visit 13: 9-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 13: 9-months Post-SOT | 11.16 |
  Visit 14: 12-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 14: 12-months Post-SOT | 11.14 |

10. Secondary Outcome: Function (i.e., Physical Recovery)
Description: The Western Ontario and McMaster University Osteoarthritis Index (WOMAC) questionnaire consists of 24 items that evaluate pain, stiffness, and physical functional disability. Each item is scored on an 11-point numerical rating scale from 0 to 10, where higher scores indicate greater pain, stiffness, and disability. For each participant, the scores from each of the 24 items were averaged to calculate the participant's total score, with a minimum score of 0 and a maximum score of 10. The mean total score was then calculated across participants and percent reduction was calculated for each time point. To be considered a success, participants must have experienced ≥ 33% reduction in their score. The number of successes is presented.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: participants (with imputed values)
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
participants (with imputed values)
  Visit 10: 8-weeks Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 10: 8-weeks Post-SOT | 16.00 | 11.00
  Visit 11: 3-months Post-SOT: number analyzed (Participants) | 20 | 20
  Visit 11: 3-months Post-SOT | 13.00 | 9.00
  Visit 12: 6-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 12: 6-months Post-SOT | 11.42 |
  Visit 13: 9-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 13: 9-months Post-SOT | 12.22 |
  Visit 14: 12-months Post-SOT: number analyzed (Participants) | 20 | 0
  Visit 14: 12-months Post-SOT | 11.08 |

11. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The total distance that a participant could walk in 6 minutes was recorded, and participants unable to walk at all were given a score of 0 meters. The mean distance was then determined across participants. The baseline score was compared to the score at the specified intervals after start of therapy.
Time Frame: Baseline (Visit 1), 8-weeks post-start of treatment (SOT) (Visit 10), and 3-months post-SOT (Visit 11)
Population: Full Analysis set presented. Data were unavailable for two Group 1 participants and one Group 2 participant at 8-weeks post-SOT and for four Group 1 participants and one Group 2 participant at 3-months post-SOT.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group 1 (Treatment) | Group 2 (Control)
Number analyzed (Participants) | 20 | 21
meters
  Visit 1: Baseline | 267.29 (108.91) | 291.94 (91.12)
  Visit 10: 8-weeks Post-SOT: number analyzed (Participants) | 18 | 20
  Visit 10: 8-weeks Post-SOT | 354.29 (197.63) | 253.36 (142.77)
  Visit 11: 3-months Post-SOT: number analyzed (Participants) | 16 | 20
  Visit 11: 3-months Post-SOT | 318.11 (164.83) | 269.77 (156.50)

ADVERSE EVENTS:
Time Frame: Each participant enrolled was assessed for adverse events from the time of informed consent through their final study visit. For Group 1, the total assessment period was approximately 13 months for each participant. Each Group 2 participant that did not crossover to receive stimulation treatment was assessed through their study participation (approximately 3 months). Group 2 participants that crossed over to receive treatment were each assessed for approximately 16 months.
Arm/Group | Group 1 (Treatment) | Group 2 (Control) | Group 2 Crossover Safety Set
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/11
Other Adverse Events (participants affected / at risk) | 9/28 | 14/27 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Treatment) (N=28) | Group 2 (Control) (N=27) | Group 2 Crossover Safety Set (N=11)
Skin irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 11 (15) | 4 (5)
Itching at bandage, pad, and/or lead exit sites (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 2 (2)
Discoloration/bruising at lead exit site (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Skin tear at bandage or connector site (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Granuloma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Unable to determine relationship to study
Exacerbation of existing pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Uncomfortable stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain at lead site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04341948/Prot_004.pdf
  • Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT04341948/SAP_005.pdf